CLINICAL TRIAL: NCT03239093
Title: Sixteen Years Trends in Reported Undernutrition in Switzerland
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Pedro Marques-Vidal, Associate professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 1
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Malnutrition; Epidemiology
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Observational study using official data from the Federal Office of Statistics

SUMMARY:
To assess 16-year trends in undernutrition reporting and management in Switzerland

DETAILED DESCRIPTION:
Analysis of data from the Swiss hospital discharge databases between 1998 and 2014. The database was provided by the Swiss federal office of statistics (http://www.bfs.admin.ch); it covers 98% of public and private hospitals within Switzerland and includes all stays for each hospital.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged ≥20 years), length of hospital stay >1 day, not having any ICD-10 codes related to pregnancy, childbirth and puerperium (i.e. ICD-10 codes beginning with letter "O") as main diagnosis, and having complete demographic data and information on main diagnosis and mortality

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalizations representing 98% of public and private hospitals within Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 13297188 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-29 (Actual); Study Completion 2017-07-29 (Actual)

PRIMARY OUTCOMES:
undernutrition reporting | 1998-2014
  ICD-10 codes E12 (undernutrition-related diabetes mellitus), E40 (kwashiorkor), E41 (nutritional marasmus), E42 (marasmic kwashiorkor), E43 (unspecified severe protein-energy undernutrition), E44 (protein-energy undernutrition of moderate and mild degree), E46 (unspecified protein-energy undernutrition), R63 (R63.0: Anorexia, R63.3: feeding difficulties and mismanagement; R63.4: abnormal weight loss and R63.6: Insufficient intake of food and water due to self-neglect), and R64 (cachexia).

SECONDARY OUTCOMES:
nutritional management | 1998-2014
  CHOP codes related to enteral nutrition (96.6 and 96.35), parenteral nutrition (99.15), nutritional advice and therapy (89.0A.30, 89.0A.31 or 89.0A.32, depending on year) and multimodal nutritional therapy (89.0A.4*, where *=any number).

OTHER OUTCOMES:
Length of stay | 1998-2014
  Overall length of hospital stay, in days
In-hospital mortality | 1998-2014
  Hospital mortality (code=deceased)
Nosocomial infection | 1998-2014
  ICD-10 codes T80.2 (Infections following infusion, transfusion and therapeutic injection); T82.6 (Infection and inflammatory reaction due to cardiac valve prosthesis); T82.7 (Infection and inflammatory reaction due to other cardiac and vascular devices, implants and grafts); T83.5 (Infection and inflammatory reaction due to prosthetic device, implant and graft in urinary system); T83.6 (Infection and inflammatory reaction due to prosthetic device, implant and graft in genital tract); T84.5 (Infection and inflammatory reaction due to internal joint prosthesis); T84.6 (Infection and inflammatory reaction due to internal fixation device [any site]); T84.7 (Infection and inflammatory reaction due to other internal orthopaedic prosthetic devices, implants and grafts); T85.7 (Infection and inflammatory reaction due to other internal prosthetic devices, implants and grafts); A04.7 (Clostridium difficile infection);

IPD SHARING:
Plan to Share IPD: No
Data request must be sent to the Swiss Federal Office of Statistics (http://www.bfs.admin.ch) and must comply with Swiss data protection rules